CLINICAL TRIAL: NCT03718702
Title: The Effectiveness of an Electronic Pain Management Programme (ePain) for Working Population With Chronic Pain: A Randomized Controlled Trial
Brief Title: The Effectiveness of an Electronic Pain Management Programme (ePain) for Working Population With Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Mun Yee Mimi, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: ePain
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Working population; Online learning
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Self-efficacy theory of behavioral change is adopted to guide the conceptual framework and development of the intervention. It was first introduced by Bandura in 1977. In the theory, self-efficacy would increase when a person participates actively in the activities to gain experience. There are two expectations in the model. The efficacy expectations of the person would contribute to the person's behaviour. The person performs the behaviour and would expect the outcomes and this is outcome expectations. The theory has been discussed for how to apply in health promotion. As the theory integrates self-efficacy and self-regulatory elements, people are benefited from the improved health outcomes which is resulted from the health behaviours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): ePain will be accessible by the intervention group.
  Interventions: Other: ePain
- Control group (No Intervention): No intervention will be applied to control group and they can download an educational pamphlet only.

INTERVENTIONS:
Other: ePain — Electronic pain management programme (ePain)
  Arms: Intervention group

SUMMARY:
Pain in commonly found in working population. The working population who aged from 15 to 64 is the largest portion of population in Hong Kong. Also, the prevalence of chronic pain in this population group is high. The issue requires special attention. Researches demonstrated pain affects a person in a multidimensional way. Pain induces negative effects to both the physical and psychological aspects. The levels of depression, anxiety, stress are increased and quality of life is decreased in people with chronic pain. They are interrelated to pain. As pain induced discomforts, people adopted self-initiated treatments as treatment. Pharmacological and non-pharmacological pain management interventions are commonly used. Although people used different ways to relieve the pain, they tend to bear the pain to work or take sick leave. This contributes to the work loss to the whole society.

Pain service in Hong Kong is scarce in the public and private sectors. It takes months for a pain sufferer to be arranged for a pain clinic follow-up. It is possible for the pain get worsen while waiting for the pain service. The pain can be difficult to treat afterwards. As self-initiated treatments are welcomed by the pain sufferers, pain education can be focused on empowering the pain sufferers on their pain knowledge and self-management techniques. The pain self-efficacy can be enhanced. The pain sufferers can be benefited from lowering the pain intensity and negative emotions. It can be a solution to develop an online pain management programme to ease the service demand.

Limited studies are found for online pain management programmes to improve the pain self-efficacy and self-management techniques. In order to fill the knowledge gap and service gap, the present study aims to evaluate an online pain management programme (ePain) in improving the self-efficacy, reduction of pain intensity, decreased levels of depression, anxiety and stress, and improving quality of life in pain management in adults with chronic pain. Participants are randomised to the intervention group or the control group.

DETAILED DESCRIPTION:
Participants will register in ePain for an individual account. Then they will finish the the pre-test questionnaire. They will be randomized to either the intervention group or control group. ePain will be accessed by the participants in the intervention group. The control group will remain their regular activities. The participants in both groups will need to complete the pre-test (Week 1), process evaluation (Week 3), post-assessment (Week 6) and follow-up assessment (Week 12). Same questionnaire will be used in the assessments. Demographic data will be collected in Week 1. At Week 1, 3, 6 and 12, pain situation and pain self-efficacy will be collected. Data of negative emotions and quality of life will be collected at Week 1, 6 and 12. The control group will undergo the same assessment as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 15 to 65;
* Performed a formal job during the seven days before the intervention or worked for pay or profit during the seven days before the intervention;
* Able to read and understand traditional Chinese;
* With non-cancer chronic pain for at least three months;
* With pain scored one or above in the numeric rating scale from zero to ten in the Chinese version of Brief Pain Inventory (BPI-C)

Exclusion Criteria:

* Adults aged 15 below or above 65;
* Not performed any formal jobs for pay or profit during the seven days before the intervention;
* With cancer pain or non-cancer acute pain for less than 3 months.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Pain self-efficacy | Baseline, Week 3, Week 6 and Week 12
  Changes from baseline to Week 3, Week 6 and Week 12 in pain self-efficacy using the Pain Self-Efficacy Questionnaire

SECONDARY OUTCOMES:
Pain situations | Baseline, Week 3, Week 6 and Week 12
  Changes from baseline to Week 3, Week 6 and Week 12 in pain situations using the Chinese version of Brief Pain Inventory (BPI-C)
Negative emotions | Baseline, Week 6 and Week 12
  Changes from baseline to Week 6 and Week 12 in depression, anxiety and stress levels using the Depression Anxiety Stress Scale (DASS-21)
Changes in level of quality of life | Baseline, Week 6 and Week 12
  Changes from baseline to Week 6 and Week 12 in quality of life using the World Health Organization Quality of Life Instruments (WHOQOL-BREF)
Feedback | Week 6
  Open ended questions developed by the research team to collect comments of using ePain, including the user experience, webpage design, usefulness of ePain and items for improvement

CONTACTS AND LOCATIONS:
Overall Officials: Mimi Tse, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, Hung Hom, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang SK, Tse MMY, Leung SF, Fotis T. The effectiveness of an electronic pain management programme for the working population with chronic pain: study protocol for a randomized controlled trial. Trials. 2020 May 24;21(1):421. doi: 10.1186/s13063-020-04348-5. PMID 32448387